CLINICAL TRIAL: NCT06059560
Title: An Open, Real-world Study of the Effects of Perioperative Intensive Nutritional Management on Short-term Quality of Life and Long-term Life Outcomes in Patients With Multiple Cancers
Brief Title: Nutritional Intervention for Patients With Multiple Cancer Types
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Kai Li, Deputy Director of surgical Oncology, First Hospital of China Medical University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FirstHCMU_nutrient
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Cancer
Keywords: nutrition; prognosis
MeSH Terms: conditions — Neoplasms | interventions — Nutrition Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventian group (Experimental): Intensive nutritional interventions based on real-world treatments
  Interventions: Dietary Supplement: Nutritional therapy
- control group (Experimental): Nutritional guidance and education based on real world treatments
  Interventions: Dietary Supplement: Nutritional therapy

INTERVENTIONS:
Dietary Supplement: Nutritional therapy — Intensive nutritional therapy based on real world therapy

SUMMARY:
To evaluate the nutritional status of patients with different types of tumors by continuous nutritional intervention and follow-up intervention in the perioperative period,and the impact on progression-free survival/survival and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* ① Age ≥18 years old, <80 years old, male or female; ② The patient signed the informed consent and volunteered to participate in the study; ③ Patients with malignant tumors (laryngeal cancer, esophageal cancer, lung cancer, gastric cancer, colorectal cancer, liver cancer, pancreatic cancer) evaluated by clinical stage II to IV; ④ Patients undergoing tumor surgery; ⑤ Patients with NRS 2002 score ≥ 3 after management risk screening; ⑥ Basic reading and communication skills; ⑦ Have the ability to act; Patients with a life expectancy greater than 6 months;

Exclusion Criteria:

* ① Acute onset of chronic disease; ② Pregnant or lactating women; ③ Patients with contraindications and no tumor surgery; (4) Patients with malignant tumors (laryngeal cancer, esophageal cancer, lung cancer, stomach cancer, colorectal cancer, liver cancer, pancreatic cancer) were confirmed by pathology and/or cytology after surgery; ⑤ Combined with cognitive dysfunction, mental disorder, consciousness disorder or unwillingness to cooperate; ⑥ Patients with severe gastrointestinal symptoms, liver and renal insufficiency (alanine aminotransferase ALT≥2 times the upper limit of normal value; Total bilirubin Tbil≥2 times the upper limit of normal value; Creatinine Cr≥2 times the upper limit of normal value); (7) Patients with two or more types of tumors; Long-term bed rest, hemiplegia or coma; ⑨ Severe dysfunction of liver, kidney and other organs; ⑩ Allergy or intolerance to nutrients or their main components (such as lactose or galactose, etc.).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Survival index | 3 years
  DFS/OS

SECONDARY OUTCOMES:
Quality of life index | 3years
  Perioperative survival index of patients with multiple cancer types

CONTACTS AND LOCATIONS:
Overall Officials: Kai Li, MD, Study Director — First Hospital of China Medical University
Locations (1):
- The First Affiliated Hospital of China Medical University, Shenyang, Liaoning, China